CLINICAL TRIAL: NCT02536014
Title: Effect of Dexmedetomidine on Heart-rate Corrected QT(QTc) Interval Prolongation During Robotic-assisted Laparoscopic Radical Prostatectomy -Randomized Blind Clinical Trial-
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 4-2015-0337
Record Dates: First submitted 2015-07-14; First posted 2015-08-31 (Estimated); Last update posted 2016-01-29 (Estimated); Status verified 2016-01

CONDITIONS: Prostate Cancer; Robotic Surgery
Keywords: Dexmedetomidine; pneumoperitoneum; trendelenburg position; QTc interval; Tp-e interval; robotic prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms; Pneumoperitoneum | interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dexmedetomidine (Experimental)
  Interventions: Drug: Dexmedetomidine
- Saline (Active Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine infusion (0.3㎍/kg/hr) from anesthetic induction to the end of pneumoperitoneum
  Arms: Dexmedetomidine
Drug: Saline — Saline infusion during the same time period
  Arms: Saline

SUMMARY:
Sympathetic activity could be increased during robot-assisted laparoscopic radical prostatectomy, which is performed in a steep trendelenburg position under CO2 pneumoperitoneum.

Stimulation of the sympathetic nervous system prolongs the QT interval and can increases the susceptibility to life threatening cardiac arrhythmias.

Dexmedetomidine has sympatholytic effects and potential antiarrhythmic properties. Perioperative administration of dexmedetomidine is a potential preventive and treatment strategy for tachyarrhythmia. Thus the investigators decided to evaluate the effect of dexmedetomidine on heart-rate corrected QT interval during robot-assisted laparoscopic radical prostatectomy. Furthermore, the investigators evaluated the Tp-e, Tp-e/QT ratio and Tp-e/QTc ratio as well.

ELIGIBILITY:
Inclusion Criteria:

1. ASA class I-II
2. Otaining written informed consent from the patients who were undergoing robot- assisted laparoscopic radical prostatectomy

Exclusion Criteria:

1. Emergency operation
2. Cardiac disease (unstable angina, congestive heart failure, valvular heart disease)
3. Ventricular conduction abnormality
4. Prior pacemaker insertion
5. Abnormal electrolyte values
6. Patients who take antiarrythmic agent
7. Hepatic or renal failure
8. Drug hyperactivity
9. Neurological or psychiatric illnesses

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-08; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Dexmedetomidine on heart-rate corrected QT(QTc) interval | From pre-induciton until 60 min after the end of pneumoperitoneum
  QTc intervals (msec) are recorded from pre-induction until 60 min after the end of pneumoperitoneum

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institue, Yonsei Universiy College of Medicine, Seoul, Seoul, South Korea